CLINICAL TRIAL: NCT04934644
Title: The Effect of Hyperbaric Oxygen Treatment in Patients With Osteoradionecrosis. A Prospective Multicenter Study.
Brief Title: The Effect of Hyperbaric Oxygen Treatment in Patients With Osteoradionecrosis.
Acronym: ORN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORN
Record Dates: First submitted 2021-05-17; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Osteoradionecrosis
Keywords: Osteoradionecrosis; Radiation injuries; Hyperbaric oxygenation; Hyperbaric oxygen treatment
MeSH Terms: conditions — Osteoradionecrosis; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen treatment (Experimental): 30 HBO treatments and standard care. If surgery is needed an additional 10 HBO treatments postoperative.
  Interventions: Procedure: Hyperbaric oxygen treatment
- Control (No Intervention): Standard care. Surgery if needed.

INTERVENTIONS:
Procedure: Hyperbaric oxygen treatment — Hyperbaric oxygen treatment 90 min from start to start of decompression. The chamber is pressurized to 2,4 ATA and the patients will be breathing 100% oxygen. Treatments will be given once daily, five days a week (no treatments on weekends and holidays).
  Arms: Hyperbaric oxygen treatment

SUMMARY:
Osteoradionecrosis (ORN) is a severe delayed radiation-induced injury that can occur in patients whom have been subjected to radiotherapy for head and neck cancer. Hyperbaric oxygen treatment (HBO) is one treatment option. In Sweden it is used in some locations in combination to standard treatment which includes for example antibiotics, pain medication and surgery. There is still not sufficient evidence that this treatment is effective in this group of patients.

The primary aim of this study will be to evaluate HBO as a treatment for osteoradionecrosis in terms of slowing the progression of the disease, or at the best, cure the disease.

DETAILED DESCRIPTION:
Radiotherapy (RT) is frequently used for treatment of head and neck cancer, in combination with surgery and chemotherapy. Although RT can improve the survival rate among head and neck-cancer patients, it has negative effects on the healthy tissue surrounding the tumour. Osteoradionecrosis (ORN) is a severe delayed radiation-induced injury that can occur in patients whom have been subjected to RT for head and neck cancer. ORN can occur within months to several years after radiotherapy. Symptoms can include pain, dysesthesia, halitosis (bad breath) exposed necrotic bone, infection, orocutaneous fistula and pathologic fractures. The mandible is the most common site affected by ORN, but other bones can be affected as well. ORN has earlier been treated with long-term antibiotics and surgery. Today the treatment is multidisciplinary and also includes local wound care, hyperbaric oxygen (HBO) and new medications for example Pentoxifylline, a vasodilator that also inhibits fibrosis, Tocopherol (Vitamin E), that reduces damage by free radicals, and Clodronate, a bisphosphonate that inhibits bone resorption.

Hyperbaric oxygen treatment (HBO) is an intervention in which the individual breathes near 100% oxygen intermittently while inside a hyperbaric chamber that is pressurized to above sea level pressure. By increasing the inspired partial pressure of oxygen (PO₂), with an increased O₂ fraction inspired and increased pressure, the amount of oxygen in blood can be increased. This also increases the distance that oxygen can diffuse from the capillaries into the tissues. HBO increase production of reactive oxygen and nitrogen species. This leads to neovascularisation by two processes: blood vessel growth by local endothelial cells (angiogenesis) and recruitment and differentiation of stem cells to form vessels "de novo" (vasculogenesis). HBO has also been shown to stimulate fibroblast proliferation and enhances collagen synthesis.

The primary aim of this study will be to evaluate HBO as a treatment for osteoradionecrosis in terms of slowing the progression of the disease, or at the best, cure the disease. As secondary aims for this study, the effect of HBO on pain, infection, mouth-opening capacity and quality of life will be evaluated.

The study will be a prospective study with matched controls evaluating the effect of HBO in comparison to standard care in patients with ORN stage 1-2b according to classification of Kagan and Schwartz. A total of 60 patients in each group will be included, which should be sufficient for statistical significance according to power calculations.

The patients will be enrolled into two groups. The first group of patients will receive HBO treatment. The treatment will be given in a multi or monoplace chamber pressurized to 2,4-2,5 ATA, 90 minutes from start to decompression, and the patients will be breathing 100 % oxygen. Treatment will be given once daily, five days a week. All patients will receive 30 treatments and if surgery is needed the patient will receive an additional 10 treatments postoperatively. All according to local routines for treatment of ORN with HBO. The control group will consist of a group of patients with the same diagnosis and same stage of ORN. These will be patients from a maxillofacial unit in Sweden not using HBO treatment or patients who decline the treatment. The controls will be matched based on sex, age, tumour-stage and RT. These patients will be treated with standard care and be subjected to surgery if needed.

Baseline visit will include clinical examination by an oral and maxillofacial surgeon and quality of life questionnaires developed and validated for head-and-neck cancer patients (EORTC QLQ C30 and H&N35). The patients in the HBO group will also be examined by a doctor at the hyperbaric unit. Follow-up will be performed every third month during the first year. In total the patients will be followed for a period of four years, every sixth months the second and third year and then on a yearly basis from the third year and on if no need for more frequent controls exist. The follow-up will include clinical examination by an oral and maxillofacial surgeon, radiographies including CT-scan and quality of life questionnaires. This is according to established care program. Blood samples, and if the patient undergoes surgery, tissue samples, will also be collected to look at biomarkers for inflammation and bone turnover.

Primary end-point of the study is changes in the bone as well as the soft tissue surrounding the necrotic bone. Secondary end-points are improvements regarding pain, infection, mouth-opening capacity and quality of life scorings.

ELIGIBILITY:
Inclusion Criteria:

* Osteoradionecrosis in the head and neck area (Stage 1-2b according to the classification by Schwartz and Kagan)
* Previous radiation with or without chemotherapy of a histologically verified primary tumor in the head and neck area.
* Patient free of tumor.
* Autonomous patient.
* Age ≥18 years old.
* WHO performance status 0-3.
* Ability to understand Swedish speech and writing.
* Received oral and written information about the study and given consent to participate in writing.

Exclusion Criteria:

* Contraindications against HBO.
* Participation in other ongoing study on osteoradionecrosis.
* Pregnancy or planned pregnancy.
* Woman in fertile age without effective contraceptive method.
* Alcohol or drug abuse.
* WHO performance status 4.
* Suspicion of recurrent tumor.
* Mental health disorder or other condition which makes the patient unable to follow study protocol.
* Not able to give informed concent.
* Previous HBO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-03-19 (Estimated); Study Completion 2024-03-19 (Estimated)

PRIMARY OUTCOMES:
SH-index | 1-4 years
  Assessment of healing of soft and hard tissue using SH-index S0H0-S1H3, where lower scores are a better outcome and higher scores are worse. The classification is based on clinical examination of the soft tissue (S) and radiographies of the hard tissue (H).

SECONDARY OUTCOMES:
Change in stage of osteoradionecrosis | 1-4 years
  Schwartz and Kagan 1a-3b, where 1 is a better outcome and 3b is worse.
Infection | 1-4 years
  3-grade scale
Transcutaneous perfusion measurement | 1-4 years
  Perfusion of blood in the affected area
Perceived pain | 1-4 years
  Visual Analog Scale (VAS) 0-10, where 0 is a better outcome an 10 is worse.
Mouth opening capacity | 1-4
  mm
Secretion of saliva | 1-4 years
  ml/min
Perceived quality of life | 1-4 years
  EORTC (European organisation for research and treatment of cancer) quality of life questionnaire (QLQ C-30). A system for evaluating quality of life in cancer patients. Score 0-100, where a higher value is a higher quality of life.
Perceived quality of life | 1-4 years
  EORTC (European organisation for research and treatment of cancer) quality of life questionnaire (QLQ H&N35). A system for evaluating quality of life in patients with head and neck cancer. Score 0-100, where a higher value means more symptoms.
Alkaline phosphatase | 1-4 years
  An increased value indicates an increase in bone metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Göran Kjeller, Docent, Study Director — Department of oral and maxillofacial surgery, Institute of odontology, Sahlgrenska Academy, GU
Locations (2):
- Sweden (2):
  - Department of oral and maxillofacial surgery, Institute of odontology, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Göteborg
  - Department of Oral and Maxillofacial Surgery, The University Hospital of Skåne, Lund, Skåne County

IPD SHARING:
Plan to Share IPD: No